CLINICAL TRIAL: NCT02193360
Title: A Phase I/II, Open Label, Multicenter, Pilot Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacodynamics of FFP104 in Subjects Previously Diagnosed With Primary Biliary Cirrhosis (PBC)
Brief Title: Pilot Study of FFP104 Dose Escalation in PBC Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fast Forward Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFP104-001; 2014-001638-27 (EudraCT Number)
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Inflammation; PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm Dose Escalation (Experimental)
  Interventions: Drug: FFP104

INTERVENTIONS:
Drug: FFP104 — Cohorts receiving multiple weekly or biweekly i.v. doses of FFP104. FFP104 dose levels: 1.0, 2.5 and 5.0 mg/kg. Subjects will be treated for 12 weeks and then followed for safety and efficacy assessments for an additional 12 weeks.

SUMMARY:
The purpose of this study is to determine the initial safety, tolerability and pharmacodynamics of the CD40-antagonist Mab, FFP104, in subjects with PBC

ELIGIBILITY:
Inclusion Criteria:

* Male or female Age between 18 and 75 years of age inclusive at the time of signing the informed consent
* Established diagnosis of PBC according to the EASL criteria (European Association for the Study of the Liver 2009): A diagnosis of PBC can be made with confidence in adult patients with otherwise unexplained elevation of ALP and presence of anti-mitochondrial antibody (AMA≥1:40), and/or AMA type M2. A liver biopsy is not essential for the diagnosis of PBC in these patients, but allows activity and stage of the disease to be assessed.
* Having a screening ALP serum level between 1.67 and 5x ULN inclusive.
* Be on a stable dose of ursodeoxycholic acid (UDCA) 12-20 mg/kg/day for at least 3 months prior to Screening or intolerant of UDCA in the opinion of the investigator (no UDCA for at least 8 weeks prior to Screening).
* Are not pregnant or breast feeding and do not plan to become pregnant or father a child during the study. Female subjects (of childbearing potential) must be willing to use two medically accepted forms of contraception throughout the study and must be willing to submit to pregnancy test(s). Male subjects must agree to use medically accepted contraception methods with their partners throughout the study as described above, unless they have had a prior vasectomy.
* Has the ability to communicate adequately with the study staff and to comply with the requirements of the entire study, with the help of a caregiver, if applicable.

Exclusion Criteria:

* Laboratory screening results

  * alanine transaminase (ALT) >5x ULN
  * aspartate transaminase (AST) >5x ULN
  * Total bilirubin >2x ULN. Isolated bilirubin >2x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%
  * Total white blood cells (WBC) <3000 cells/mm3
  * Absolute neutrophil count (ANC) <1500 cells/mm3
  * Platelet count <100,000/mm3
  * Prothrombin time (international normalized ratio (INR)> 1.2
* Body mass index (BMI) ≥35 or suspected to have relevant nonalcoholic fatty liver disease (NAFLD) as based on the judgment of the Investigator at screening
* Subject has a history of, or current viral hepatitis B or C (including hepatitis B surface antigen [HBsAg], hepatitis B core antibody and hepatitis C virus (HCV) antibody [anti-HCV] positivity), or a positive HIV antibody screen at time of screening
* Recipients of liver or other organ transplantation or anticipated need for orthotropic organ transplantation in one year as determined by the Mayo Risk Score
* Co-existing liver or biliary diseases, such as primary sclerosing cholangitis, choledocholithiasis, acute or chronic hepatitis, autoimmune hepatitis, alcoholic liver disease, nonalcoholic steatohepatitis (NASH), acute infection of bile duct system or gall bladder, history of gastrointestinal bleeding (secondary to portal hypertension), cholangiocarcinoma diagnosed or suspected liver cancers
* Recurrent variceal hemorrhage, uncontrolled encephalopathy, Child-Pugh Class B/C, Esophageal Varices, or refractory ascites within the previous 6 months of Screening (defined as date informed consent signed)
* Have a family history (more than one first degree relative) of multiple thrombotic events or a personal history of any venous or arterial thrombotic event including deep vein thrombosis, stroke, myocardial infarction, pulmonary embolus, or peripheral arterial thromboembolic events
* Prohibited medications 6 months prior to Screening: azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate mofetil, pentoxifylline; fenofibrate or other fibrates; budesonide and other systemic corticosteroids; potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazid, or nitrofurantoin)
* Prohibited medications 12 months prior to Screening: antibodies or immunotherapy directed against interleukins or other cytokines or chemokines
* Subjects with recurrent bacterial infections (as judged by the Investigator) within 6 months prior to first dose of FFP104, active bacterial, fungal or mycobacterial infections observed during screening, or any recent episode of infection requiring hospitalizations or treatment with antibiotics (within the 3 months prior to first dose)
* History of malignancy, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ
* Immunization with a live vaccine within 4 weeks of Screening with the exception of influenza vaccine and no planned immunisations within the period of the study
* Known clinically significant cardiac disease (e.g., myocardial infarction or stroke, unstable angina, claudication, etc.), or evidence of a clinically significant electrocardiogram (ECG) abnormality within the previous 12 months prior to Screening
* Subjects with evidence of other serious, significant, acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study
* History of recent (within 12 months of study) alcohol or drug abuse
* Use of other immunosuppressive medications 4 weeks prior to Screening
* Active tuberculosis (TB) in the past or currently suspected TB which is presently receiving treatment or prophylactic therapy, has a positive TB test (as defined by local biological requirements), or any significant abnormality on chest X-ray within 3 months prior to Screening
* Subjects who have planned surgery during the study period or have undergone major surgery within the 3 months prior to Screening
* Known clinically significant allergy or known hypersensitivity to drugs that, in the opinion of the Investigator, may affect the patient's safety
* Known sensitivity to any component of the study drug or previous sensitivity reaction or other clinically significant reaction to intravenous medications or biologic therapy
* Participated to another clinical trial within the past 30 days prior to Screening, or is still within a washout period of a previous clinical trial or has previously received FFP104 (PG102) or ch5D12 in this or any study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of FFP104 in PBC subjects following repeat doses of FFP104 | Days 1, 3, 5 and weeks 2 - 12, 14, 16 and 24
  Safety outcomes include abbreviated physical examination, treatment emergent adverse events (TEAE), clinically significant changes in clinical haematology, clinical chemistry, and urinalysis.

SECONDARY OUTCOMES:
Proportion of subjects with a 10% decrease in Alkaline Phosphatase (ALP) from baseline values | Week 12
Proportion of subjects with a 25 and 40% decrease in ALP from baseline | Weeks 4, 8 and 12
Proportion of subjects with ALP<1.67 from upper limit of normal (ULN), an ALP decrease >15% and bilirubin within normal levels | Weeks 4, 8, 12 and 24
Proportion of subjects with a biochemical response according to 'Paris I' criteria: ALP≤ 3x ULN and Aspartate Transaminase (AST) ≤2x ULN and bilirubin ≤1mg/dL | Weeks 4, 8, 12 and 24
To evaluate the individual and mean changes in serum liver biochemistry from baseline | Weeks 2, 4, 8, 12, 16 and 24
  Evaluation of individual and mean changes in lab values (serum ALP, AST, bilirubin, albumin and gamma glutamyl transpeptidase (GGT)) over time from baseline values
To evaluate changes from baseline with Mayo Risk Score | Weeks 4, 8, 12 and 24
To evaluate changes from baseline in the Patient Report Outcome PBC-40 Quality of Life | Weeks 12 and 24
To evaluate changes from baseline in pruritus using the Visual Analog Scale (VAS) | Weeks 12 and 24
To evaluate changes from baseline in fatigue using the VAS | Weeks 12 and 24
To evaluate changes in serum FFP104 levels from baseline | over time

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (2):
  - Amsterdam Medical Center, Amsterdam
  - Erasmus University Medical Center, Rotterdam
- United Kingdom (3):
  - University Hospital Birmingham, Birmingham
  - Royal Free Hospital, London
  - Newcastle upon Tyne Hospitals, Newcastle upon Tyne